CLINICAL TRIAL: NCT05708313
Title: Effects of 9-18 Weeks of Intensive Cardiac Rehabilitation After a Major Cardiovascular Event in Patients With Cardiovascular Disease-AHH-ICR
Brief Title: Effects of 9-18 Weeks of Intensive Cardiac Rehabilitation After a Major Cardiovascular Event in Patients With CVD
Acronym: AHH-ICR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AHH-002
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cardiovascular Diseases; Lifestyle Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Groups will be assigned to the exercise treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Rehabilitation (Experimental): people recruited for the trial will participate in the Intensive cardiac rehabilitation arm.
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Behavioral: lifestyle modification — Participants will undergo an exercise program designed by AHH
  Other Names: exercise

SUMMARY:
Implement an intensive cardiac rehabilitation program at Arkansas Heart Hospital (AHH) to find out if the AHH-ICR is equivalent to the CMS approved programs when it comes to results.

DETAILED DESCRIPTION:
Implement the ICR Program to determine if

1. AHH-ICR will increase patients physical and psychological well-being and is non-superior/comparable to current ICR programs.
2. To determine the most appropriate ICR program protocols to improve fitness and decrease cardiovascular risk factors.
3. To determine if the ICR program has a direct relationship to improvements in the health of cardiovascular patients.
4. To determine non-inferiority to already established ICR programs in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for cardiac rehab per CMS requirements.
2. Males and Females Age ≥ 65≤ 85 years
3. Acute myocardial infarction within the preceding 6 months
4. Coronary artery bypass surgery
5. Current stable angina pectoris (chest pain)
6. Heart valve repair or replacement
7. Percutaneous transluminal coronary angioplasty or coronary stenting
8. BMI ≥ 18 ≤35
9. HgA1C ≤10

Exclusion Criteria:

- 1. Renal or hepatic dysfunction 2. Amputees (unless both groups have similar patients) 3. Current chemo/radiation treatment (unless both groups have similar patients) 4. Malnutrition 5. HIV/AIDS 6. Post-Bariatric surgery patients 7. History of substance abuse 8. Gastroparesis 9. Patients taking Warfarin/Coumadin 10. CHF patients on fluid restrictions requiring monitoring of water intake from food and liquids.

11. Cognitive deficits that would preclude cardiac rehabilitation 12. Patients with physical limitations that would prevent cardiac rehabilitation 13. Patients who are unable to attend the program 14. Patient who live >45… miles from cardiac rehab center

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 198 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Serum Lipid | Baseline to program completion (9-18 weeks)
  Total cholesterol, ADH, LDL and triglycerides (mg/dl)
Body Mass Index | Baseline to program completion (9-18 weeks)
  calculated from Height and weight.
Resting Blood Pressure | Baseline to program completion (9-18 weeks)
  Systolic and Diastolic Blood Pressure (mmHg)
Hemoglobin A1c | Baseline to program completion (9-18 weeks)
  measure in whole blood (normal 4.5-6.2 (%))

SECONDARY OUTCOMES:
Dartmouth Coop quality of Life Questionnaire | Baseline to program completion (9-18 weeks)
  Self-Reported assessment of participant general health
Hospital Re-admission rate | Baseline to program completion (9-18 weeks)
  Number of time patient is admitted to the hospital for cardiovascular related events.
Patient Health Questionnaire (PHQ9) | Baseline to program completion (9-18 weeks)
  Assessment of perceive depression state.
Duke Activity Index | Baseline to program completion (9-18 weeks)
  Assessment of physical Activity
6-minute walk test | Baseline and at program completion (9-18 weeks)
  Distance walked in 6 minutes (mts)
Medication Changes | Baseline to program completion (9-18 weeks)
  decrease medications intake..
Perceived Exertion (RPE) | Baseline to program completion (9-18 weeks)
  as perceived by patient in the Rating of perceived Exertion scale.
Resting Metabolic Rate | Baseline to program completion (9-18 weeks)
  measure in Kcal using the Mifflin-St. Jeor equation.
Diet intake | Baseline to program completion (9-18 weeks)
  food records using the Passio App.

CONTACTS AND LOCATIONS:
Overall Officials: Leybi Ramirez Kelly, Study Director — Arkansas Heart Hospital/Arkansas Site Management Services LLC
Locations (1):
- Arkansas Heart Hospital-Clinic, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be share with other investigators outside of the research facility unless is for data analysis and publication

REFERENCES:
- [Background] Bethell HJ. Cardiac rehabilitation: from Hellerstein to the millennium. Int J Clin Pract. 2000 Mar;54(2):92-7. PMID 10824363
- [Background] 3. Cardiac Rehabilitation Updated: Oct 31, 2018 Author: Vibhuti N Singh, MD, MPH, FACC, FSCAI; Chief Editor: Consuelo T Lorenzo, MD
- [Background] Razavi M, Fournier S, Shepard DS, Ritter G, Strickler GK, Stason WB. Effects of lifestyle modification programs on cardiac risk factors. PLoS One. 2014 Dec 9;9(12):e114772. doi: 10.1371/journal.pone.0114772. eCollection 2014. PMID 25490202
- [Background] Hill J, Timmis A. Exercise tolerance testing. BMJ. 2002 May 4;324(7345):1084-7. doi: 10.1136/bmj.324.7345.1084. No abstract available. PMID 11991917
- [Background] American College of Sports Medicine Position Stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 1998 Jun;30(6):992-1008. PMID 9624662
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Wenger NK, Froelicher ES, Smith LK, Ades PA, Berra K, Blumenthal JA, Certo CM, Dattilo AM, Davis D, DeBusk RF, et al. Cardiac rehabilitation as secondary prevention. Agency for Health Care Policy and Research and National Heart, Lung, and Blood Institute. Clin Pract Guidel Quick Ref Guide Clin. 1995 Oct;(17):1-23. PMID 8595435
- [Background] Kothmann E, Batterham AM, Owen SJ, Turley AJ, Cheesman M, Parry A, Danjoux G. Effect of short-term exercise training on aerobic fitness in patients with abdominal aortic aneurysms: a pilot study. Br J Anaesth. 2009 Oct;103(4):505-10. doi: 10.1093/bja/aep205. Epub 2009 Jul 23. PMID 19628486
- [Background] Rosenfeldt F, Braun L, Spitzer O, Bradley S, Shepherd J, Bailey M, van der Merwe J, Leong JY, Esmore D. Physical conditioning and mental stress reduction--a randomised trial in patients undergoing cardiac surgery. BMC Complement Altern Med. 2011 Mar 9;11:20. doi: 10.1186/1472-6882-11-20. PMID 21385466
- [Background] Sawatzky JA, Kehler DS, Ready AE, Lerner N, Boreskie S, Lamont D, Luchik D, Arora RC, Duhamel TA. Prehabilitation program for elective coronary artery bypass graft surgery patients: a pilot randomized controlled study. Clin Rehabil. 2014 Jul;28(7):648-57. doi: 10.1177/0269215513516475. Epub 2014 Jan 23. PMID 24459173
- [Background] Hadj A, Esmore D, Rowland M, Pepe S, Schneider L, Lewin J, Rosenfeldt F. Pre-operative preparation for cardiac surgery utilising a combination of metabolic, physical and mental therapy. Heart Lung Circ. 2006 Jun;15(3):172-81. doi: 10.1016/j.hlc.2006.01.008. Epub 2006 May 19. PMID 16713353
- See also: Equipment used — https://www.gehealthcare.com